CLINICAL TRIAL: NCT02049437
Title: AIDS 347: IL-6 Blockade in Treated HIV Infection
Acronym: IL-6
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AIDS 347; IL-6 (Other Grant/Funding Number: U01-AI-105937-01)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: HIV; Immune failure; Tocilizumab; ACTEMRA; Antiretroviral therapy; HAART
MeSH Terms: conditions — HIV Infections | interventions — tocilizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: TCZ, then placebo (Active Comparator): ARM A: TCZ, 4 mg/Kg by IV infusion over 60 minutes (not to exceed 400 mg) once at study entry, followed by TCZ, 8 mg/Kg by IV infusion over 60 minutes (not to exceed 800 mg) at weeks 4 and 8, and THEN placebo by IV infusion at weeks 20, 24, and 28.
  Interventions: Drug: tocilizumab; Drug: Placebo
- Arm B: Placebo, then TCZ (Placebo Comparator): ARM B: Placebo by IV infusion at study entry followed by placebo by IV infusion at weeks 4 and 8, and THEN TCZ, 4 mg/Kg (not to exceed 400 mg) by IV infusion over 60 minutes once at week 20, followed by TCZ, 8 mg/Kg (not to exceed 800 mg) by IV infusion over 60 minutes at weeks 24 and 28.
  Interventions: Drug: tocilizumab; Drug: Placebo

INTERVENTIONS:
Drug: tocilizumab — Subjects will be randomized 1:1 to one of the following arms:
  ARM A: TCZ, 4 mg/Kg by IV infusion over 60 minutes (not to exceed 400 mg) once at study entry, followed by TCZ, 8 mg/Kg by IV infusion over 60 minutes (not to exceed 800 mg) at weeks 4 and 8, and THEN placebo by IV infusion at weeks 20, 24, and 28.
  ARM B: Placebo by IV infusion at study entry followed by placebo by IV infusion at weeks 4 and 8, and THEN TCZ, 4 mg/Kg (not to exceed 400 mg) by IV infusion over 60 minutes once at week 20, followed by TCZ, 8 mg/Kg (not to exceed 800 mg) by IV infusion over 60 minutes at weeks 24 and 28.
  Other Names: TCZ
Drug: Placebo — Subjects will be randomized 1:1 to one of the following arms:
  ARM A: TCZ, 4 mg/Kg by IV infusion over 60 minutes (not to exceed 400 mg) once at study entry, followed by TCZ, 8 mg/Kg by IV infusion over 60 minutes (not to exceed 800 mg) at weeks 4 aned 8, and THEN placebo by IV infusion at weeks 20, 24, and 28.
  ARM B: Placebo by IV infusion at study entry followed by placebo by IV infusion at weeks 4 and 8, and THEN TCZ, 4 mg/Kg (not to exceed 400 mg) by IV infusion over 60 minutes once at week 20, followed by TCZ, 8 mg/Kg (not to exceed 800 mg) by IV infusion over 60 minutes at weeks 24 and 28.
  Other Names: Normal saline for infusion

SUMMARY:
The study is a phase I/II, double-blind, placebo-controlled, randomized cross-over clinical trial of tocilizumab (TCZ) or placebo in HIV-infected subjects receiving antiretroviral therapy with suppressed viral replication and CD4+ T cell count ≥350 and ≤1,000 cells/mm3)

DETAILED DESCRIPTION:
DESIGN The study is a phase I/II, double-blind, placebo-controlled, randomized cross-over clinical trial of tocilizumab (TCZ) or placebo in HIV-infected subjects receiving antiretroviral therapy with suppressed viral replication and CD4+ T cell count ≥350 and ≤1,000 cells/mm3)

DURATION 40 weeks during cross-over treatment periods total per subject.

SAMPLE SIZE 30 subjects with complete data up to week 30. Up to 36 subjects may be enrolled in order to achieve an estimated final sample size of 30 participants with complete data up to week 30.

POPULATION HIV-infected male and female subjects from 18 through 60 years of age receiving combination antiretroviral therapy (ART) without changes in the 24 weeks prior to enrollment (changes for reasons other than virologic failure allowed up to 8 weeks prior to enrollment), with a suppressed plasma HIV RNA (<200 copies/mL, one blip up to <1,000 copies/mL permitted) for at least 96 weeks and a CD4+ T-cell count ≥350 and ≤1,000 cells/mm3 at the time of study enrollment.

REGIMEN Subjects will be randomized 1:1 to one of the following arms:

ARM A: TCZ, 4 mg/Kg by IV infusion over 60 minutes (not to exceed 400 mg) once at study entry, followed by TCZ, 8 mg/Kg by IV infusion over 60 minutes (not to exceed 800 mg) at weeks 4, and 8 and THEN placebo by IV infusion at weeks 20, 24, and 28.

ARM B: Placebo by IV infusion at study entry followed by placebo by IV infusion at weeks 4 and 8, and THEN TCZ, 4 mg/Kg (not to exceed 400 mg) by IV infusion over 60 minutes once at week 24, followed by TCZ, 8 mg/Kg (not to exceed 800 mg) by IV infusion over 60 minutes at weeks 24 and 28.

ELIGIBILITY:
Inclusion Criteria

4.1.1 Men and women age 18-60 years.

4.1.2 Ability and willingness to communicate in English or Spanish

4.1.3 Ability and willingness of subject to provide informed consent.

4.1.4 Ability and willingness to provide adequate locator information.

4.1.5 HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test at any time before study entry and confirmed by a licensed Western blot, a second antibody test by a method other than rapid HIV or E/CIA; HIV-1 antigen; or plasma HIV-1 RNA viral load.

4.1.6 Receiving a stable antiretroviral regimen consisting of 3 or more drugs belonging to two or more classes, one of which must be a protease inhibitor, an integrase inhibitor, or a non-nucleoside reverse transcriptase inhibitor, without any changes due to virologic failure in the past 24 weeks, and with no plans to change antiretroviral regimen in the 40 weeks following enrollment. If the regimen includes a protease inhibitor, ritonavir or an approved boosting agent known to increase trough levels of the protease inhibitor by at least 50% must also be a part of the regimen.

NOTE A: Changes to the antiretroviral regimen 8 weeks or more prior to enrollment are allowed if the plasma HIV RNA was <50 copies/mL at the time of the change, the reason for the change was not suspicion or documentation of virologic failure, and all other criteria for virologic control, as outlined in criterion 4.1.9 below, are met.

NOTE B: For the purposes of this protocol, "a change due to virologic failure" is defined as any of the following events or combinations thereof happening in a patient who is receiving uninterrupted combination antiretroviral therapy including at least three agents belonging to at least two classes: a) plasma HIV RNA is >200 copies/mL on two or more consecutive occasions; b) the treating physician determines that any given plasma HIV RNA value is indicative or suggestive of virologic failure, and recommends that the patient's regimen be modified as a result; c) a genotypic or phenotypic antiretroviral resistance test identifies the presence of resistance to any component of a patient's regimen that was not present before, and a physician recommends that the patient's regimen be modified as a result.

4.1.7 For subjects who have a positive HBcAb only:

• An antiretroviral regimen containing one or more of the following medications: lamivudine, emtricitabine, or tenofovir.

4.1.8 Screening CD4+ T-cell count ≥350 cells/mm3 but ≤1,000 cells/mm3 performed in a laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.

4.1.9 HIV-1 RNA <200 copies/mL at every time a plasma HIV RNA has been obtained, but no fewer than twice, in the 96 weeks prior to enrollment.

NOTE: One plasma HIV RNA above 200 copies/mL but lower than 1,000 copies in the 96 weeks prior to enrollment is permissible if flanked by two measurements that are both below 200 copies. The HIV-1 RNA at screening must be <50 copies/mL.

4.1.10 The following laboratory values obtained within 60 days prior to entry:

* Hgb ≥10 g/dL
* Platelet count >100,000/mm3
* Absolute neutrophil count (ANC) ≥2,000 cells/mm3
* Aspartate aminotransferase (AST) [serum glutamic oxaloacetic transaminase (SGOT)] <1.5x ULN
* Alanine aminotransferase (ALT) [serum glutamic pyruvic transaminase (SGPT)] <1.5x ULN
* For subjects who consent to undergo rectal tissue sampling only: International normalized ratio (INR) < 1.7
* Total bilirubin <3.0 mg/dL, EXCEPT for subjects receiving atazanavir
* For subjects receiving atazanavir: Direct bilirubin ≤1.0 mg/dL
* Calculated GFR ≥60 mL/min/1.73m2

4.1.11 Female subjects of reproductive potential must have a negative serum or urine pregnancy test at study entry and must affirm that they do not intend to become pregnant for the duration of the study.

NOTE: For the purposes of this protocol, a female subject of reproductive potential is defined as one who has reached menarche, has not been post-menopausal for at least 24 consecutive months (i.e., has had menses within the preceding 24 months), and has not undergone surgical sterilization (e.g., hysterectomy, tubal ligation, or bilateral oophorectomy).

4.1.12 Female subjects of reproductive potential participating in sexual activity that could lead to pregnancy must agree to use at least one of the following forms of birth control for at least 30 days prior to study entry through 30 days after the final study visit:

* Condoms (male or female) with or without a spermicidal agent
* Diaphragm or cervical cap with spermicide

PLUS at least one of the following:

* An FDA-approved copper intrauterine device (IUD), e.g. ParaGard®, or an FDA-approved hormone-releasing IUD, e.g. Mirena®
* An FDA-approved transdermal hormonal contraceptive, e.g. Ortho-Evra®
* An FDA-approved injectable hormonal contraceptive, e.g. Depo-Provera®
* An FDA-approved hormonal contraceptive in vaginal ring form, e.g. NuvaRing®
* An FDA-approved implantable hormonal contraceptive, e.g. Implanon® or Jadelle®

NOTE A: Oral hormonal contraceptives, either combined or progestin-only, are not acceptable as a second contraceptive method.

NOTE B: Women of reproductive potential who are using a hormonal contraceptive not included above may consider switching their contraceptive to one of the approved forms, but will be required to do so in consultation with their primary healthcare providers. Study investigators will not prescribe or recommend a specific form of contraception to study participants. The study will not cover the costs of contraceptives.

4.1.13 Female subjects who are not of reproductive potential [i.e., women who have been post-menopausal for at least 24 consecutive months or women who have undergone surgical sterilization (e.g., hysterectomy, tubal ligation, or bilateral oophorectomy)] are eligible without requiring the use of a contraceptive. Acceptable documentation of sterilization, other contraception methods, menopause and reproductive potential is patient-reported history at any time prior to screening.

4.1.14 Subjects must be determined by the investigators to have at least one fully active regimen available to them other than the regimen they are receiving at study entry. The determination of whether or not an alternative regimen is available must take into account both the subject's antiretroviral history and any previously obtained resistance testing. A valid alternative regimen must meet the recommendations for an active regimen outlined in the current DHHS guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents (93).

Exclusion Criteria

4.2.1 History of one of the following opportunistic infections at any time in the past, as demonstrated by either a patient-reported or physician-documented diagnosis AND the initiation of specific treatment if applicable:

* Tuberculosis, pulmonary or extrapulmonary
* Non-tuberculous mycobacterial infection, disseminated or extrapulmonary
* Pneumocystis jirovecii pneumonia
* Coccidioidomycosis, disseminated or extrapulmonary
* Cryptococcosis, extrapulmonary
* Cryptosporidiosis or isosporiasis, chronic intestinal (greater than 1 month's duration)
* Cytomegalovirus disease (other than liver, spleen, or lymph nodes) and including retinitis with loss of vision
* Histoplasmosis, disseminated or extrapulmonary
* Kaposi's sarcoma
* Lymphoma, Burkitt's or immunoblastic, regardless of anatomical location
* Lymphoma, primary of brain
* Progressive multifocal leukoencephalopathy
* Toxoplasmosis of brain

4.2.2 Latent tuberculosis infection, defined as a positive or borderline FDA-approved interferon-gamma release assay (IGRA).

4.2.3 Pregnant or breastfeeding.

4.2.4 Active local or systemic infection (defined as requiring systemic antibiotics or other medical or surgical treatment) at the time of enrollment.

4.2.5 Use of systemic cancer chemotherapy or radiation therapy, immunosuppressive or immunomodulatory therapy (e.g., interferons, tumor necrosis factor antagonists, interleukins) or any investigational therapy within 90 days prior to study entry or continued indication for such medications. A list of prohibited study medications is provided in appendix 1 of the Manual of Operations (MOPS).

NOTE A: Use of inhaled or nasal steroids, the equivalent of 10 mg of prednisone or less per day or a less than 2-week course of steroids are not exclusionary.

NOTE B: A single course of 1% hydrocortisone cream or equivalent applied up to 3 times a day to <10 square inches area for <2 weeks is permitted. The investigators will determine if other forms of limited, short-term topical steroid use are expected to interfere significantly with the study objectives and are therefore exclusionary.

4.2.6 Receipt of a live attenuated vaccine within 30 days prior to study entry or expected need for such vaccines at any time during and for 30 days after the study.

4.2.7 Known allergy/sensitivity or any hypersensitivity to components of the study drug or its formulation.

4.2.8 Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

4.2.9 Serious illness requiring systemic treatment and/or hospitalization within 45 days prior to study entry.

4.2.11 Known cirrhosis or severe liver disease (e.g., ascites, encephalopathy, history of variceal bleeding).

4.2.12 Active hepatitis B (positive HBsAg, HBV DNA, or HBeAg) or hepatitis C (positive HCV antibody and positive HCV RNA in plasma) documented at the screening visit.

NOTE A: For purposes of documenting hepatitis B status, an HBsAg or HBV DNA obtained in the 6 months prior to and up to the date of the screening visit is acceptable EXCEPT for subjects with a positive HBcAb at screening (see Note B). A negative HBeAg during the same period in the absence of an HBsAg or HBV DNA is not sufficient evidence of HBV-negative status. If a clinically obtained test is not available at screening, an HBsAg will be drawn together with other evaluations at this visit.

NOTE B: For subjects with a positive HBcAb at screening, an HBV DNA below the limit of quantification at any time from screening to study entry is required.

NOTE C: For purposes of documenting HCV status, a negative HCV antibody obtained in the 6 months prior to and up to the date of the screening visit is sufficient. For any subject with a positive HCV antibody, an HCV RNA measurement is required.

4.2.13 History of diverticulitis, intestinal perforation, distal intestinal obstruction, or lower gastrointestinal bleeding.

4.2.14 An antiretroviral regimen containing maraviroc at study entry. 4.215 History of a demyelinating disorder such as multiple sclerosis or chronic demyelinating polyneuropathy at any time in the past.

4.2.16 A trough level of any protease inhibitor (other than a boosting dose of ritonavir) or non-nucleoside reverse transcriptase inhibitor included in the subject's antiretroviral regimen at screening that is below the lower limit of the steady-state trough level range observed in published studies, according to Table 2, below.

Table 2: Cutoffs of selected antiretroviral trough levels Drug Lower limit of range (levels below this at screening are exclusionary) Efavirenz(94) 1 µg/mL Nevirapine(94) 3 µg/mL Etravirine(95) 75 ng/mL Rilpivirine(96) 4 ng/mL Atazanavir/r(94) 0.15 µg/mL Darunavir/r(96) 1036 ng/mL Lopinavir/r(94)

1 µg/mL Amprenavir(94) 0.4 µg/mL Fosamprenavir/r(94) 0.4 µg/mL Indinavir/r(94) 0.1 µg/mL Saquinavir SGC/r(94) 0.1 µg/mL Nelfinavir(94) 0.8 µg/mL

4.2.17 Active malignant disease, other than a resected basal cell carcinoma of the skin.

4.2.18 For subjects who consent to undergo rectal tissue sampling only:

* History of a bleeding diathesis of any kind, or contraindication for lower GI endoscopy
* Major GI tract surgery within 45 days prior to study entry. Minor procedures involving only the anal canal such as condyloma ablations, hemorrhoidectomy, and anoscopy are permitted if cleared by the responsible surgeon.
* Continued need for, or use during the 7 days prior to the scheduled flex-sig procedure, of the following medications:

  * Aspirin, systemic antiplatelet agents, or more than 4 doses of NSAIDs
  * Warfarin, heparin, thrombin inhibitors, factor Xa inhibitors, and systemic thromobolytics and fibrinolytics. A list of prohibited medications for the flex-sig procedure can be found in the appendix of the MOPS. A bridge course of short-acting low-molecular weight heparin within the 7-day pre-procedure window in patients receiving a chronic systemic anticoagulant who can be safely maintained off anticoagulation for several days is permitted if cleared by the subject's primary healthcare provider and the UHCMC Digestive Health Institute.
* Abnormalities of the colorectal mucosa, or significant colorectal symptoms, which in the opinion of the clinician represent a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benigno Rodriguez, MD, Study Chair — Case Western Reserve University; Michael Lederman, MD, Study Chair — Case Western Reserve University; George Yendewa, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Clinical Research Site, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Funderburg NT, Shive CL, Chen Z, Tatsuoka C, Bowman ER, Longenecker CT, McComsey GA, Clagett BM, Dorazio D, Freeman ML, Sieg SF, Moisi D, Anthony DD, Jacobson JM, Stein SL, Calabrese LH, Landay A, Flexner C, Crawford KW, Capparelli EV, Rodriguez B, Lederman MM. Interleukin 6 Blockade With Tocilizumab Diminishes Indices of Inflammation That Are Linked to Mortality in Treated Human Immunodeficiency Virus Infection. Clin Infect Dis. 2023 Jul 26;77(2):272-279. doi: 10.1093/cid/ciad199. PMID 37011013

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Placebo, Then TCZ: ARM B: Placebo by IV infusion at study entry, followed by placebo by IV infusion at weeks 4 and 8, and THEN TCZ, 4 mg/Kg (not to exceed 400 mg) by IV infusion over 60 min once at week 20, followed by TCZ, 8 mg/Kg (not to exceed 800 mg) by IV infusion over 60 min at weeks 24 and 28.
Period: Period 1
Arm/Group | Arm A: TCZ, Then Placebo | Arm B: Placebo, Then TCZ
Started | 17 | 17
Completed | 15 | 16 (Dropout due to low trough levels)
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Adverse Event | 1 | 0
Period: Washout 1
Arm/Group | Arm A: TCZ, Then Placebo | Arm B: Placebo, Then TCZ
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Arm A: TCZ, Then Placebo | Arm B: Placebo, Then TCZ
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Washout 2
Arm/Group | Arm A: TCZ, Then Placebo | Arm B: Placebo, Then TCZ
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: TCZ, Then Placebo | Arm B: Placebo, Then TCZ | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [42 to 53] | 49 [44 to 54] | 48 [42 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 10 | 17
  Black or African American | 10 | 6 | 16
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 2 or Greater AEs
Description: The number and percentage of participants experiencing at least one grade ≥2 clinical or laboratory adverse event related to study treatment during each period (0 to 10 weeks for Period 1 or 20 to 30 weeks for Period 2).
Time Frame: 30 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Tocilizumab: Patients from Arm A that obtained TCZ, 4 mg/kg by IV infusion over 60 min (not to exceed 400 mg) once at study entry, followed by TCZ, 8 mg/kg by IV infusion over 60 min (not to exceed 800 mg) at weeks 4, and 8.
  Patients from Arm B that obtained TCZ, 4 mg/kg by IV infusion over 60 min (not to exceed 400 mg) once at week 20, followed by TCZ, 8 mg/kg (not to exceed 800 mg) by IV infusion over 60 minutes at weeks 24 and 28 after the first (placebo) interventional period and washout period
- Placebo: Patients from Arm A that, after washout period 1, obtained placebo by IV infusion at weeks 20, 24 and 28.
  Patients from Arm B that obtained placebo by IV infusion at study entry followed by placebo by IV infusion at weeks 4 and 8.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 10 | 2
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.07, Mixed Models Analysis; Risk Ratio (RR) = 4.43, 95% CI 2-sided [0.90 to 21.83]

2. Secondary Outcome: Serum C-reactive Protein Change Between Beginning and End of Treatment Period
Description: The primary analysis of the two co-primary (CRP and T cell cycling) endpoints will specifically focus on the changes from study entry to week 10 and from week 20 to week 30.
Time Frame: study entry - 10 weeks; 20 weeks - 30 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 31 | 31
ng/mL
  Serum C-reactive protein at either study entry or week 20 | 4316 (6907) | 3320 (4149)
  Serum C-reactive protein at either 10 weeks or 30 weeks | 157 (183) | 2256 (1928)
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -2036.8, 95% CI 2-sided [-3490.32 to -900.62]

3. Secondary Outcome: Change in Proportion of Central Memory T Cells Expressing Ki67 Between Beginning and End of Treatment Period
Description: as for outcome 2
Time Frame: study entry - 10 weeks; 20 weeks - 30 weeks
Measure: Mean (Standard Deviation); unit: proportion of central memory T cells
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 31 | 31
proportion of central memory T cells
  proportion of central memory T cells expressing Ki67 at either study entry or 20 weeks | 0.0689 (0.0222) | 0.0721 (0.0293)
  proportion of central memory T cells expressing Ki67 at either 10 weeks or 30 weeks | 0.0685 (0.0192) | 0.0708 (0.0222)
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.79 to 0.65]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the total length of the trial, 40 weeks.
Description: 33 patients were at risk for adverse events during the Toculizumab treatment: 17 patients in arm A that started Toculizumab in period 1 + 16 patients in arm B that started Toculizumab in period 2 32 patients were at risk for adverse events during the placebo treatment: 17 patients in arm B that started placebo in period 1 + 15 patients in arm A that started placebo treatment in period 2
Arm/Group | Tocilizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/32
Other Adverse Events (participants affected / at risk) | 23/33 | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=33) | Placebo (N=32)
Severe neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — ANC<500
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=33) | Placebo (N=32)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hidradentitis Suppurativa (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (2)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute gout flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abnormal blood test (General disorders) | 21 (45) | 15 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT02049437/Prot_SAP_000.pdf